CLINICAL TRIAL: NCT06584669
Title: Investigation of Krill Oil in Women with Premenstrual Syndrome: a Randomized, Placebo-controlled, Double-blind, Parallel Group Study with Different Dosages
Brief Title: Investigation of Krill Oil in Women with Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AKBM041H
Record Dates: First submitted 2024-08-28; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Premenstrual Syndrome
Keywords: inflammation; krill oil; omega-3 fatty acids; premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, parallel group study
Who Masked: Participant, Investigator
Masking Description: All participants and study staff were blinded to treatment allocations until the last patient had completed the last visit. The study capsules were identical in shape and color and packed in blisters tailor-made for each intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 0.5 KO (Active Comparator): This group receives 500 mg Krill Oil + 1.5 g medium-chain triglycerides (MCT) Oil daily during a 4-cycle supplementation phase.
  Interventions: Dietary Supplement: Krill oil
- 1 KO (Active Comparator): This group receives 1 g Krill Oil + 1 g MCT Oil daily during a 4-cycle supplementation phase.
  Interventions: Dietary Supplement: Krill oil
- 2 KO (Active Comparator): This group receives 2 g Krill Oil daily during a 4-cycle supplementation phase.
  Interventions: Dietary Supplement: Krill oil
- 0.5 KO+A (Active Comparator): This group receives 500 mg Krill Oil + 2mg astaxanthin + 1.5 g MCT Oil daily during a 4-cycle supplementation phase.
  Interventions: Dietary Supplement: Krill oil
- Placebo (Placebo Comparator): This group receives medium-chain triglyceride (MCT) oil daily during a 4-cycle supplementation phase.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Krill oil — The krill oil capsules contain Superba™ krill oil extracted from Antarctic krill (Euphausia superba).
  Arms: 0.5 KO; 0.5 KO+A; 1 KO; 2 KO
Other: Placebo — The placebo capsules contain a medium-chain triglyceride (MCT) oil obtained by fractionation of coconut and palm kernel oil, which has no detectable levels of EPA, DHA, astaxanthin, or phospholipids.
  Arms: Placebo

SUMMARY:
In this study the effects of different dosages and preparations of krill oil in comparison to placebo on symptoms of premenstrual syndrome in healthy, female adults will be assessed.

DETAILED DESCRIPTION:
The study is a randomized, placebo-controlled, double-blind, parallel group trial, in which the effect of krill oil is investigated in healthy female volunteers showing premenstrual symptoms. The study period covers a time period over 6 menstrual cycles of women under which the first two cycles are recorded to assess baseline conditions followed by a 4-cycle supplementation phase. Volunteers are randomly allocated to the 5 study groups including placebo and 4 different dosages and formulations of krill oil. Over the whole study period, volunteers report daily their symptoms in the validated questionnaire DRSP. Mood state and quality of life are assessed at baseline and after two and 4 cycles of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Age: 20 - 50 years
* Sex: female
* Premenopausal
* Regular menstrual bleeding
* History of and presence of PMS symptoms of at least 6 months
* Subject is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry, haematology

Exclusion Criteria:

* BMI: < 19 kg/m2, ≥ 30 kg/m2
* Heavy smoker >15 cigarettes / day
* Known pregnancy, breast feeding or intention to become pregnant during the course of the study
* No use of acceptable contraceptive method during the study
* Menstrual cycle lasting less than 24 / longer than 35 days
* Hormone treatment because of premenstrual symptoms
* Diagnosed premenstrual dysphoric disorder (PMDD), a severe form of PMS
* Regular consumption of omega-3 fatty acids (e.g. nutritional supplements) within previous 3 months or during the study course
* Fish consumption of more than 1 serving of fatty fish (e.g herring, mackerel, salmon) per week
* Relevant allergy or known hypersensitivity against compounds of the study preparations
* Unstable medical illness or relevant history or presence of any medical disorder, potentially interfering with this study (e.g. volunteers having experienced any cardiovascular events such as infarction, angina, surgical endocoronary intervention, stroke in the last 6 months or psychiatric disorders / psychoactive medication)
* Clinically relevant abnormal laboratory, ECG, vital signs or physical findings at screening
* Intake of medication potentially interfering with this study
* Known malabsorption / maldigestion
* Drug-, alcohol- and medication abuses
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 2 weeks prior to study start (day 1) or during study
* Participation in any other clinical study within the last 30 days prior to study start or during the study
* Any other condition that, based on Investigator's judgement, makes the subject unfit for inclusion into study
* Anticipating any planned changes in lifestyle for the duration of the study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2013-04-11 (Actual); Study Completion 2013-08-23 (Actual)

PRIMARY OUTCOMES:
Measurement of reduction in premenstrual symptoms in the late luteal phase | Daily from baseline to study completion, up to 6 months
  Reduction in premenstrual symptoms in the late luteal phase, as measured by the Daily Record of Severity of Problems (DRSP), following supplementation with 2 g krill oil compared to placebo. All other products are assessed as secondary outcomes.

SECONDARY OUTCOMES:
Measurement of total DRSP score in mid follicular phase | Daily from baseline to study completion, up to 6 months
  Measures the overall severity of symptoms using the Daily Rating of Severity of Problems (DRSP) scale during the mid-follicular phase. It combines daily ratings to reflect symptom intensity for this specific phase.
Measurement of physical Items Subscore | Daily from baseline to study completion, for up to 6 months
  The Physical Items Subscore assesses the severity and frequency of physical symptoms experienced by participants, such as fatigue, headaches, and muscle pain. These symptoms are evaluated daily using a standardized scale, where each symptom is rated based on intensity and impact on daily functioning. The scores in scale points are combined to create a subscore representing the overall physical symptom burden.
Measurement of mood Items Subscore | Daily from baseline to study completion, up to 6 months
  This subscore assesses the severity of mood-related symptoms, such as anxiety and irritability, rated daily on a standardized scale. Scores in scale points reflect the overall emotional symptom burden.
Measurement of physical Items Subscore | Daily from baseline to study completion, for up to 6 months.
  The Physical Items Subscore assesses the severity and frequency of physical symptoms experienced by participants, such as fatigue, headaches, and muscle pain. These symptoms are evaluated daily using a standardized scale, where each symptom is rated based on intensity and impact on daily functioning. The scores in scale points are then combined to create a subscore representing the overall physical symptom burden.
Measurement of total Score on Q-LES-Q SF | Daily from baseline to study completion, up to 6 months
  Evaluates overall quality of life using the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q SF). This score reflects the combined daily assessments of various life satisfaction and enjoyment domains given in scale points.
Measurement of quantity of analgesics consumed | Daily from baseline to study completion, up to 6 months
  Tracks the number of analgesic doses taken daily by participants. This measure reflects the overall usage of pain relief medication throughout the study.
Measurement of total mood disturbance score on POMS | Daily from baseline to study completion, for up to 6 months
  Assesses the overall mood disturbance using the Profile of Mood States (POMS) scale. This score given in scale points combines daily ratings to indicate the intensity of mood disturbances experienced by participants.
Measurement of proportion of responders with 50% reduction in late luteal phase symptoms | Daily from baseline to study completion, up to 6 months
  Measures the percentage of participants who show a 50% reduction in symptoms during the late luteal phase. This reflects the effectiveness of the intervention in alleviating symptoms during this phase.
Measurement of Omega-3 Index | Baseline and at 6 months post-intervention
  Assesses the Omega-3 Index by measuring the percentage of EPA and DHA in red blood cells. This reflects the level of Omega-3 fatty acids, indicating dietary intake and compliance.
Measurement of global assessment score at visits 4 and 6 | At 4 and 6 months
  Evaluates overall health and symptom severity during study visits 4 and 6 using a standardized scale. This score reflects participants' general condition at these specific time points.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, PhD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: Undecided